CLINICAL TRIAL: NCT06432179
Title: Pathways to Hospice Volunteering: a Grounded Theory Study
Brief Title: Hospice Volunteer Community，Dying Patient Prepare Spirtal Care
Acronym: volunteer
Status: Active, not recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202303083RINC
Record Dates: First submitted 2023-05-01; First posted 2024-05-29 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-04

CONDITIONS: Hospital Acquired Condition
Keywords: hospice Volunteer
MeSH Terms: conditions — Iatrogenic Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- hospice volunteer: Pathways to hospice volunteering: a grounded theory study

SUMMARY:
Due to the aging population, the cases of elderly disability and death caused by chronic diseases and cancer are also increasing; thus increasing the demand and trend of community palliative care. Anning volunteers are members of the Anning team and play an integral role in the care of the "whole community". Partners who can provide psychosocial support in fear, grief, informal care, and "individualized care" can focus on patient and family needs and give their time and presence. And make up for the shortage of medical manpower. Assist nurses to take care of patients together, which is an important support for nursing care. In the community, An Ning volunteers are an important help to closely care for patients and support family members to take care of them at home and fulfill their wish of dying at home. In view of the community's peaceful home care, the trend and importance of hospice at home, it is necessary to cooperate with the "volunteers" of the tranquility team. Inquiry Only a few papers mentioned Anning volunteers' service history and research on the meaning of life, but there was a lack of in-depth and systematic discussions on Anning volunteers, including their motivation, training, process, care effectiveness, impact on training volunteer organization management, and volunteer retention. Therefore, the motivation of the research was aroused, and it was hoped to use grounded theory to explore the motivation and process of becoming an Anning volunteer, and to identify related concepts, and finally establish a theoretical framework to describe the relevant decision-making mentality. Also serves as a reference for volunteer organization management training and retention of palliative care volunteers.

DETAILED DESCRIPTION:
The purpose of this study is to use grounded theory to explore the motivation and process of becoming a tranquility volunteer, identify relevant concepts, and finally establish a theoretical framework to describe the relevant decision-making process.

This study adopts semi-structured in-depth interviews and semi-structured one-on-one interviews to collect data. During the interview process, according to the actual situation, the interview questions will be flexibly fine-tuned according to the data analysis results.

The data coding of grounded theory is divided into three levels: open decoding, axial decoding and selective decoding; through these three levels of coding, the data are decomposed, compared, conceptualized and integrated, and finally a theory is formed.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 or above (2) Community hospice volunteers, who have served for more than one year (including one year), are currently serving volunteers or have stopped serving volunteers (3) Can speak Mandarin or Taiwanese communicate.

Exclusion Criteria:

* Those who could not understand or conduct the interview due to any physical or psychological or cognitive factors were excluded.
* no Dmentia stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — men and women
Study Population: Community hospice volunteers
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-04-29 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathways to hospice volunteering: a grounded theory study bason interview interview The 60-minute in week 24 | base on week 24
  Using qualitative research to interview volunteers' motivations, journeys and training processes as volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Chun Tang, PHD, Principal Investigator — professer
Locations (1):
- Nation Taiwan university hospictal, Taipei County, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Possibility to give back to training institution results